CLINICAL TRIAL: NCT03285685
Title: Effect of Noninvasive Neuromodulation on Chronic Pain and Anxiety Levels in Individuals With Temporomandibular Disorders
Brief Title: Effect of Noninvasive Neuromodulation on Chronic Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Tatyanne dos Santos Falcão Silva, Tatyanne Falcão, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NeuroDTM
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Temporomandibular Dysfunction (TMD)
Keywords: Analgesia; Facial pain; Transcranial Direct Current Stimulation; Temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Agnosia; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS M1 (Experimental): active tDCS Participants will receive active transcranial direct current stimulation.
  Interventions: Device: active tDCS
- tDCS DLPF (Experimental): active tDCS Participants will receive active transcranial direct current stimulation.
  Interventions: Device: active tDCS
- tDCS sham (Sham Comparator): tDCS Sham Participants will receive sham transcranial direct current stimulation.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — Duration: 20 minutes; Intensity: 2 mA; Placement: anodal over left M1 and cathodal over supraorbital contralateral area
  Arms: tDCS M1
Device: active tDCS — Duration: 20 minutes; Intensity: 2 mA; Placement: anodal over left DLPFC and cathodal over supraorbital contralateral area.
  Arms: tDCS DLPF
Device: sham tDCS — The procedure is the same as for active tDCS anodal over left M1 and cathodal over supraorbital contralateral area, but the in the placebo tDCS the stimulation is non-active / sham.
  Arms: tDCS sham

SUMMARY:
1. BACKGROUND: Temporomandibular Dysfunction (TMD) is a disease characterized by a set of signs and symptoms that may include joint noise, pain in the mastication muscles, limitation of mandibular movements, facial pain, joint pain and / or dental wear. Pain appears as a very present and striking symptom, with a tendency to chronicity. This is a difficult treatment condition often associated with psychological factors such as anxiety. Chronic pain involved modifications in the neuronal excitability, therefore, the neuromodulation withTranscranial direct current stimulation (tDCS) appears as a possible strategy for the treatment. Some studies have shown improvement in subjects with chronic pain using tDCS, however, it needs further investigation of its therapeutic effect.
2. PROBLEM: Despite the wide range of strategies used to treat patients with TMD, some patients have a temporary and / or unsatisfactory relief response, which generates hypotheses that emotional components often underlie treatment refractoriness, and development of a memory for pain. Thus, it is evident the need for a therapy that acts directly on the central nervous system (CNS). This action can occur through medications, however, many individuals are refractory or have side effects such as dependence and / or tolerance. In this way, the importance of new treatments involving neuromodulation and neuroplasticity mechanisms, such as tDCS, is highlighted, which may become a complementary alternative to the different types of treatment already in use. Besides corroborating with the need to give preference to reversible and non-invasive procedures.
3. HYPOTHESIS: The investigators believe that the use of anodic tDCS in the treatment of patients with TMD presenting with chronic pain will have a positive effect, promoting a decrease in painful symptoms through a Central Nervous System (neuromodulation) action in comparison to placebo stimulation. Because of the mutual influence between pain and psychological factors, it is expected that the analgesic effect will have a positive effect on anxiety levels. In addition, it is believed that a more intense analgesic effect occurs in the DLPF stimulation group of the cortex compared to the M1 stimulation group, since this region demonstrates to be responsible for the processing of the emotional component of the pain, often underlying the refractoriness to treatment
4. AIM: To evaluate and compare the efficacy of anodic tDCS, applied in different cortical regions (M1 and DLPFC), in the pain and anxiety levels in individuals with chronic pain due muscular TMD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years, both male and female
* Provide informed consent to participate in the study;
* Having a diagnosis of muscular pain DTM according to IA and IB, axis I RDC/TMD
* Visual analogic scale (VAS) score from 4 to 10 for six months or longer
* Presence of moderate depressive symptoms through SCL-90 scale evaluation of Axis II, (RDC / TMD)
* Not pregnant;
* Not have contraindications to tDCS, such as metal implants on the head or implanted brain devices;
* Not have history of alcohol or drugs abuse within the past 6 months as self-reported
* Not use of carbamazepine within the past 6 months as self reported
* Not have any history of epilepsy, stroke, moderate-to-severe traumatic brain injury or severe migraines
* Not have history of neurosurgery as self-reported
* Not have history of major psychiatric disorders such as schizophrenia and bipolar disorder
* Not have any other previously diagnosed disorder with symptoms similar to the DTM, such as fibromyalgia.

Exclusion Criteria:

* Two absences during treatment sessions;
* During the research, go against some criteria of inclusion mentioned above, as in the case of women, getting pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10-02 (Estimated); Primary Completion 2018-01-26 (Estimated); Study Completion 2018-02-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogic Scale | 4 months
  The visual analogic scale allows us to convert subjective sensations as pain on numerical data. A 10cm scale where 0cm is no pain and 10cm the worse imaginable pain, will be used and the subjects will be asked to mark a point on the scale representing their pain. This instrument will be used to compare the VAS values before and after the intervention.

SECONDARY OUTCOMES:
Patient Global Impression of Change Scale (PGICS) | 4 months
  The Patient Global Impression of Change Scale (PGICS) is an understandable, adequate, easy-to-use instrument capable of measuring the perception of change in health status and satisfaction with the treatment of individuals with chronic musculoskeletal pain. It is a one-dimensional measurement instrument in which individuals rate their improvement associated with intervention on a 7-item scale ranging from 1 (no change) to 7 (Much better).
State-Trait Anxiety Inventory | 4 months
  The STAI is used to evaluate objectively both aspects of anxiety: trait and state. Thus, the anxiety state will assess the level of anxiety at the specific time the test is performed and the anxiety trait will investigate the individual's willingness to react to stress situations. It is an instrument with 40 descriptive statements about the feelings of the person, distributed in two parts (trace and state of anxiety), in which each part is formed by 20 affirmations and the answers are given in scale of the type Likert of four points (1 - absolutely not the 4 - very much). The score in each questionnaire ranges from 20 to 80, with an anxiety level rating of: low (20 to 33), mean (33 to 49) and high (49 to 80).

CONTACTS AND LOCATIONS:
Locations (1):
- Tatyanne Falcão, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No